CLINICAL TRIAL: NCT02804568
Title: A Multiple-dose, Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ALKS 3831 in Adult Subjects With Schizophrenia
Brief Title: A Phase 1 Safety Study in Adults With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALK3831-A104
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Alkermes; ALK 3831; Samidorphan
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Olanzapine/samidorphan 10 mg/10 mg
  Interventions: Drug: ALKS 3831
- Group 2 (Experimental): Olanzapine/samidorphan 20 mg/10 mg
  Interventions: Drug: ALKS 3831

INTERVENTIONS:
Drug: ALKS 3831 — Oral capsule, daily administration

SUMMARY:
This study will determine the safety, tolerability, and pharmacokinetics (PK) of olanzapine and samidorphan in adults with schizophrenia following 14 consecutive days of oral administration of ALKS 3831.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) of 18.0-35.0 kg/m^2, inclusive
* Has a primary diagnosis of schizophrenia
* Capable of understanding and complying with the procedures, requirements, and restrictions of the protocol.
* Appropriate for outpatient treatment
* Agrees to abide by the contraception requirements specified in the protocol for the duration of the study or is surgically sterile
* Willing and able to provide government-issued identification
* Is in good physical health
* Agrees to maintain normal tobacco use as well as normal activities/exercise throughout the study
* Additional criteria may apply

Exclusion Criteria:

* Is currently pregnant or breastfeeding
* Initiated first antipsychotic treatment within the past 12 months, or <1 year has elapsed since the initial onset of active-phase schizophrenia symptoms
* Poses a current suicide risk at Visits 1 or 2
* Has a history of poor or inadequate response to treatment with olanzapine
* Has used a long-acting injectable antipsychotic medication in the last 6 months with the exception of 3-month paliperidone, which must not have been received within the past 12 months.
* Requires or has had electroconvulsive therapy (ECT) treatment in the 6-month period prior to Visit 1
* Has a diagnosis of alcohol or drug use disorder (with the exception of nicotine)
* Has taken opioid agonists (codeine, oxycodone, tramadol, or morphine) within the 14 days prior to Visit 1 and/or anticipates a need to take opioid medication during the study period.
* Has taken opioid antagonists including naltrexone (any formulations) and naloxone within 60 days prior to Visit 1, or has used any extended-release formulation of an opioid antagonist within 2 months prior to screening
* Tests positive for amphetamines/methamphetamine, cocaine, barbiturates, opioids (codeine, hydrocodone, hydromorphone, methadone, morphine, oxycodone, oxymorphone, and buprenorphine), phencyclidine and benzodiazepines.
* Has a known or suspected intolerance, allergy or hypersensitivity to olanzapine or opioid antagonists.
* Additional criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 15 days of dosing
Area under the concentration vs time curve over the 24 hour dosing interval (AUC0-24h) | Up to 15 days of dosing

SECONDARY OUTCOMES:
Safety will be determined by incidence of drug-related adverse events | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: David McDonnell, MD, Study Director — Alkermes, Inc.
Locations (3):
- United States (3):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Clementon, New Jersey
  - Alkermes Investigational Site, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun L, McDonnell D, von Moltke L. Pharmacokinetics and Short-term Safety of ALKS 3831, a Fixed-dose Combination of Olanzapine and Samidorphan, in Adult Subjects with Schizophrenia. Clin Ther. 2018 Nov;40(11):1845-1854.e2. doi: 10.1016/j.clinthera.2018.09.002. Epub 2018 Oct 20. PMID 30348514